CLINICAL TRIAL: NCT02934815
Title: Relational and Emotional Mechanisms of a Supportive-expressive Group Intervention (SEGT) for Women With Breast Cancer
Brief Title: Relational and Emotional Mechanisms of a Supportive-expressive Group Intervention in Breast Cancer
Acronym: BC-SEGT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Centro Hospitalar De São João, E.P.E. (Other); Mama Help - Support Centre for Breast Cancer Patients (Unknown)
Responsible Party: Principal Investigator, Tânia Brandão, Ph.D. Student, Universidade do Porto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FPCEUP/BreastCancerCare
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: psychological intervention; breast cancer; supportive-expressive group therapy; emotion regulation; social support; attachment; quality of life
MeSH Terms: conditions — Breast Neoplasms; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group - SEGT (Experimental): 16 weekly sessions, 90 min of Supportive-expressive group therapy
  Interventions: Other: Supportive-expressive group therapy
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Supportive-expressive group therapy — The supportive-expressive group therapy (SEGT) is an intervention for women with BC that is designed to build bonds and to facilitate changes in emotional expression and regulation taking into account the role that emotions play in physiologic function, intimately related to the progression of the disease. It is based on seven main themes: building bonds, expressing feelings, detoxifying dying, reordering life priorities, improve support from and communication with family and friends, fortifying families, dealing with doctors, and control pain and anxiety. Although originally developed according to an existential perspective, recently the supportive-expressive group therapy has been used according to an attachment framework.
  Other Names: SEGT
  Arms: Intervention group - SEGT

SUMMARY:
To test the feasibility of supportive-expressive group intervention (SEGT) for women with primary breast cancer and to provide a preliminary test of its efficacy.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of a 16-sessions group intervention (Supportive-Expressive group therapy) versus control group (no intervention) in women with primary breast cancer.

This study tries to evaluate the efficacy of SEGT on breast cancer patients' emotion regulation, social support, caregiving, and marital satisfaction, and its improvement on breast cancer patients' life quality. This study also intents to explore the moderating role of attachment on these associations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary breast cancer

Exclusion Criteria:

* attendance at a cancer support group or individual psychotherapy
* diagnosis of recurrent breast cancer
* severe psychiatric disorder
* history of drug or alcohol abuse

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The World Health Organization Quality of Life - BREF

SECONDARY OUTCOMES:
Change in emotion suppression across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The Emotion Regulation Questionnaire
Change in emotional self-efficacy across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The Stanford Emotional Self-Efficacy Scale-Cancer
Change in cognitive emotion across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The Cognitive Emotion Regulation Questionnaire
Change in social support across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The Multidimensional Scale of Perceived Social Support
Change in caregiving across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The Caregiving Questionnaire
Change in marital relationship across time | T0 - before the intervention; T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  Relationship Assessment Scale

OTHER OUTCOMES:
Change in group climate across time | T1 - 2 months later; T2 - 4 months later; T3 - 10 months later
  The Group Climate Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tânia Brandão, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No